CLINICAL TRIAL: NCT01176136
Title: Organizational Skills Interventions for Children With ADHD
Brief Title: Organizational Skills Interventions for Children With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0479; R305A090305 (Other Grant/Funding Number: Department of Education: Institute for Education Sciences)
Record Dates: First submitted 2010-07-12; First posted 2010-08-05 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; School-Based; Organizational Skills; Homework; Time Management
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Organizations; ALPL protein, human; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HOPS Intervention (Experimental): Middle school age children who receive the Homework, Organization, and Planning Skills (HOPS) intervention.
  Interventions: Behavioral: Homework, Organization, and Planning Skills (HOPS) Intervention
- Treatment As Usual (No Intervention): Middle school age children randomly assigned to receive treatment-as-usual services available through the school and community.

INTERVENTIONS:
Behavioral: Homework, Organization, and Planning Skills (HOPS) Intervention — HOPS is a 16 session school-based intervention. School counselors and psychologists deliver the intervention during the school day. Each session lasts 20 minutes. Initially, sessions are 2 times per week and the entire HOPS intervention is completed in 11 weeks. The study uses a waitlist control design. HOPS intervention participants (Arm 1) receive the intervention in the fall quarter of the school year and Treatment As Usual participants (Arm 2) receive the intervention in the spring quarter.
  Arms: HOPS Intervention

SUMMARY:
Attention-Deficit/Hyperactivity Disorder (ADHD) is one of the most commonly diagnosed childhood disorders, with prevalence rates estimated at 8% (Froehlich et al. 2007). Several of the primary symptoms of ADHD relate to problems with temporal and materials organization (i.e. often has difficulty organizing tasks and activities, often loses things, is often forgetful, and often fails to finish school-work, chores, or duties; APA, 2000). In the school setting, problems with organization manifest as forgetting to complete or losing homework assignments, difficulties planning for the completion of long-term projects and studying for tests, and problems keeping class materials organized. These organizational difficulties become particularly problematic in middle school and can result in considerable academic impairment (Evans, Serpell, & White, 2005). Children with ADHD underachieve academically and are more likely than their peers to receive failing grades, be retained and to drop out of school (Barkley, Fischer, Edelbrock, & Smallish, 1990).

Given the relationship between temporal and materials organization and poor school performance, it is clear there is a need for interventions to address these difficulties. We recently sought to address this need by completing a small randomized trial of an organizational skills intervention for children with ADHD (Langberg, Epstein, Urbanowicz, Simon, & Graham, (2008). The intervention was highly effective in improving materials organization and homework management and resulted in significant improvements in homework problems and grade point average. These results demonstrate the considerable promise of organizational skills interventions for children with ADHD. However, the Langberg et al. intervention was implemented as an after-school program operated by research staff with minimal involvement from school personnel. In order to promote the widespread adoption of interventions that address the organizational skills deficits of children with ADHD, the intervention must be feasible for school counselors and psychologists to implement within the time constraints of a typical school day. Accordingly, the primary goal of this study is to adapt and refine the existing intervention protocol (Langberg et al., 2008) to create a product that is highly acceptable to parents, children, teachers, school counselors and school psychologists and is feasible for school personnel to implement during the school day.

In Phase I of the proposed research, middle school counselors, psychologists, teachers, middle school students with ADHD and their parents will consult with the intervention developers to modify the after-school treatment protocol for in-school implementation. An intervention protocol will be developed. The intervention will be piloted with ten children in order to identify barriers to implementation. Measures of treatment fidelity, skills acquisition, and satisfaction will be completed. These data will inform additional modifications of the protocol and further improve feasibility/acceptability of the intervention procedures.

In Phase II of the study, school counselors/psychologists from at least four separate school districts will implement the protocol developed in Phase I. Using a waitlist control design, sixty children with ADHD in grades 6, 7, and 8 will receive the intervention. Organizational skills, grade point average, and academic impairment will be evaluated at baseline, post intervention and at 8-week follow-up. After implementing the intervention, all participants (i.e., teachers, counselors, psychologists, children and parents) will participate in a series of focus groups and will complete intervention satisfaction questionnaires. These data will inform final revisions to the intervention protocol. The resulting product will be an intervention that targets organizational skills in children with ADHD that has potential for widespread school-based dissemination. The final intervention protocol and effect size estimates from the proposed research will lay the foundation for an IES Goal III test of efficacy.

The specific aims of the project are as follows:

1. Utilize the existing organizational skills intervention protocol (Langberg et al. in press), focus group and case study data to develop an empirically and clinically informed manualized temporal and materials organization intervention for middle school children with ADHD aimed at reducing academic impairment (Phase I).
2. Refine and finalize the intervention protocol through a waitlist control trial (N=60) in a minimum of four diverse school districts, collection of clinical outcomes and completion of follow-up focus groups to assess satisfaction, feasibility, and acceptability (Phase II).

ELIGIBILITY:
Inclusion Criteria:

* Middle school age adolescents (grades 6-8) who meet Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for a diagnosis of ADHD.

Exclusion Criteria:

* Cognitive Functioning: Full scale IQ score of less than 75.
* Exclusionary Psychiatric Conditions: Students who meet diagnostic criteria for Bipolar Disorder, psychotic disorder, pervasive developmental disorders, substance dependence, or obsessive-compulsive disorder be excluded from participation.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Homework Problems Checklist | 8 months post-baseline
  Parent completed measure that assesses homework completion difficulties and homework management difficulties.

SECONDARY OUTCOMES:
Children's Organizational Skills Scales (COSS) | 8-months post-baseline
  Parent, child, and teacher completed measure that evaluates organization and time-management/planning skills.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Langberg, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States